CLINICAL TRIAL: NCT00242775
Title: Efficacy and Safety of Symbicort ®Turbuhaler® 160/4.5 µg/Inhalation, Two Inhalations Twice Daily Plus As-needed Compared With Seretide™ Diskus™ 50/500 µg/Inhalation, One Inhalation Twice Daily Plus Terbutaline Turbuhaler 0.4 mg/Inhalation As-needed - a 6-month, Randomised, Double-blind, Parallel-group, Active Controlled, Multinational Phase IIIB Study in Adult and Adolescent Patients With Persistent Asthma (AHEAD).
Brief Title: Comparison of the Efficacy/Safety of Symbicort® Turbuhaler®,Seretide™ Diskus™ 50/500 µg & Terbutaline Turbuhaler® 0.4 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5890C00002; EurodraCT No. 2004-004905-11; AHEAD
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Salmeterol Xinafoate

INTERVENTIONS:
Drug: Budesonide/formoterol Turbuhaler
  Other Names: Symbicort
Drug: Salmeterol/fluticasone Diskus

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a variable dose of Symbicort with a high fixed maintenance dose of another asthma medication, Seretide, in the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with asthma since at least 6 months prior to first visit
* Prescribed daily use of glucocorticosteroids for at least 3 months prior to first visit
* At least one asthma exacerbation more than one but less than twelve months prior to first visit

Exclusion Criteria:

* Respiratory infection affecting asthma within 30 days before first visit
* Use of oral, rectal, or parenteral glucocorticosteroids for within 30 days before first visit
* Any significant disease or disorder that may jeopardize the safety of the patient

Additional inclusion and exclusion criteria will be evaluated by the Investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2100
Dates: Start 2005-05; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of severe asthma exacerbations
Mild asthma exacerbations
FEV1
Patient-reported outcomes regarding disease status (inlc. PEF), collected via questionnaires and diaries
Healthcare utilization
Safety (adverse events)
- all variables assessed over the 6 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (143):
- Argentina (7):
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Monte Grande, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Santa Fé, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
  - Research Site, San Miguel de Tucumán
- Australia (14):
  - Research Site, Bankstown, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Bundaberg, Queensland
  - Research Site, Carina Heights, Queensland
  - Research Site, Mackay, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Toorak Gardens, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Rosebud, Victoria
  - Research Site, Nedlands, Western Australia
- Brazil (8):
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Florianópolis, Santa Catarina
  - Research Site, São Paulo, São Paulo
  - Research Site, Curitiba
  - Research Site, São Paulo
- Canada (15):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Ste-Foy, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
- China (6):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Nanjin
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Shenyang
- France (24):
  - Research Site, Angers
  - Research Site, Bernay
  - Research Site, Béthune
  - Research Site, Chamalières
  - Research Site, Férolles-Attilly
  - Research Site, Grasse
  - Research Site, Hénin-Beaumont
  - Research Site, La Rochelle
  - Research Site, Laon
  - Research Site, Le Havre
  - Research Site, Lille
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Saint-Denis
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Sélestat
  - Research Site, Toulouse
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villejuif
- Germany (21):
  - Research Site, Cottbus, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
  - Research Site, Jena-Maua, Thuringia
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Erfurt
  - Research Site, Geesthacht
  - Research Site, Großhansdorf
  - Research Site, Hagen
  - Research Site, Kassel
  - Research Site, Koblenz
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Neuruppin
  - Research Site, Sonneberg
  - Research Site, Witten
- India (4):
  - Research Site, Coimbatore
  - Research Site, Hyderbad
  - Research Site, Mumbai
  - Research Site, Noida
- Indonesia (6):
  - Research Site, Semarang, Central Java
  - Research Site, Jakarta Timur, Jakarta - Indonesia
  - Research Site, Bandung
  - Research Site, Jakarta
  - Research Site, Jakarta Timur
  - Research Site, Solo
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Seremban
- Mexico (3):
  - Research Site, Zapopan, Jalisco
  - Research Site, Villahermosa, Tabasco
  - Research Site, México
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Iloilo City
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- South Africa (15):
  - Research Site, Bryanston, Gauteng
  - Research Site, Florida Park, Gauteng
  - Research Site, Lenasia, Gauteng
  - Research Site, Linksfield, Gauteng
  - Research Site, Sandton, Gauteng
  - Research Site, Witbank, Gauteng
  - Research Site, Hillcrest, Pretoria
  - Research Site, Bellville
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Lyttelton Manor
  - Research Site, Pretoria
- Spain (11):
  - Research Site, Barcelona, Barcelona
  - Research Site, Santander, Cantabria
  - Research Site, Granada, Granada
  - Research Site, San Sebastián, Guipuzcoa
  - Research Site, Jaén, Jaén
  - Research Site, Madrid, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Seville, Sevilla
  - Research Site, Vitoria-Gasteiz, Vitoria
  - Research Site, Zaragoza, Zaragoza
  - Research Site, Seville
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
- Research Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Lin JT, Chen P, Zhou X, Sun TY, Xie CM, Xiu QY, Yao WZ, Yang L, Yin KS, Zhang YM. Budesonide/formoterol maintenance and reliever therapy in Chinese patients with asthma. Chin Med J (Engl). 2012 Sep;125(17):2994-3001. PMID 22932169
- [Derived] Bousquet J, Boulet LP, Peters MJ, Magnussen H, Quiralte J, Martinez-Aguilar NE, Carlsheimer A. Budesonide/formoterol for maintenance and relief in uncontrolled asthma vs. high-dose salmeterol/fluticasone. Respir Med. 2007 Dec;101(12):2437-46. doi: 10.1016/j.rmed.2007.07.014. Epub 2007 Oct 1. PMID 17905575